CLINICAL TRIAL: NCT02216643
Title: Randomization of Endovascular Treatment With Stent-retriever and/or Thromboaspiration vs. Best Medical Therapy in Acute Ischemic Stroke Due to Large VEssel OcclusioN Trial
Brief Title: EndoVascular Treatment With Stent-retriever and/or Thromboaspiration vs. Best Medical Therapy in Acute Ischemic Stroke
Acronym: RESILIENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Medtronic (Industry); Penumbra Inc. (Industry); iSchemaView, Inc (Unknown); Brainomix Limited (Industry)
Responsible Party: Principal Investigator, SHEILA CRISTINA OURIQUES MARTINS, MD, PHD, Stroke Neurologist, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22042613.6.1001.5327
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Ischemic Stroke
Keywords: Stroke; Ischemic Stroke; Thrombectomy; Reperfusion Therapy; Treatment
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Thrombectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thrombectomy (Experimental): mechanical thrombectomy with stentriever Solitaire FR® and/or thromboaspiration with Penumbra System® in patients with large vessel occlusion in cerebral anterior circulation vessels
  Interventions: Procedure: Thrombectomy; Device: Stentriever Solitaire FR® or Penumbra System®
- best medical treatment (No Intervention): best medical treatment in patients with acute ischemic stroke with anterior circulation large vessel occlusion

INTERVENTIONS:
Procedure: Thrombectomy — Patients with acute ischemic stroke with anterior circulation large vessel occlusion will be randomized to receive mechanical thrombectomy with stent-retriever Solitaire FR® and/or thromboaspiration with Penumbra System® versus medical management alone versus medical management alone. A maximum of six attempts to retrieve the thrombus in a single vessel can be made . No additional treatment will be allowed either with IA tPA, other mechanical devices or angioplasty/stenting.
  Other Names: Endovascular treatment; Intrarterial treatment; Endovascular revascularization
  Arms: thrombectomy
Device: Stentriever Solitaire FR® or Penumbra System® — Patients with acute ischemic stroke with anterior circulation large vessel occlusion will be randomized to receive mechanical thrombectomy with stent-retriever and/or thromboaspiration versus medical management alone versus medical management alone. A maximum of six attempts to retrieve the thrombus in a single vessel can be made . No additional treatment will be allowed either with IA tPA, other mechanical devices or angioplasty/stenting.
  Arms: thrombectomy

SUMMARY:
Prospective, multi-center, randomized, controlled, open, blinded-endpoint trial with a sequential design. The randomization employs a 1:1 ratio of mechanical thrombectomy with stentriever and/or Thromboaspiration versus medical management alone. Randomization will be done under a minimization process using age, baseline NIHSS, use of IV tpa, vessel occlusion site and hospital. To evaluate the hypothesis that mechanical thrombectomy is superior to medical management alone in achieving more favorable outcomes in the distribution of the modified Rankin Scale scores at 90 days in subjects presenting with acute large vessel ischemic stroke <8 hours from symptom onset. Subjects are either ineligible for IV alteplase or have received IV alteplase therapy without recanalization. Sample size is projected to be 690 patients for a difference in treatment effect of 10%.

DETAILED DESCRIPTION:
Patients with acute ischemic stroke related to anterior circulation large vessel occlusion will be randomized up to 8 hours from symptoms onset in both arms (mechanical thrombectomy versus medical management alone). Subjects are either ineligible for IV alteplase or have received IV alteplase therapy without recanalization. They will be admitted at acute stroke units in Brazil (or ICU if needed) and treated following international guidelines. Concomitant medications and non-pharmacological therapies will be recorded. A maximum of six attempts to retrieve the thrombus in a single vessel can be made. No additional treatment will be allowed either with Intrarterial tPA, mechanical devices or angioplasty/stenting.

The primary endpoint will be distribution of the modified Rankin Scale scores at 90 days (shift analysis) as evaluated by two separate assessors who are blinded to treatment

Interim Analysis The sample size for this Phase III Trial is projected to be 690 subjects. For interim analyses, the method of Lan and DeMets will be used to allocate alpha via the power family method with φ (phi) equal to 1 for the assessment of efficacy and futility, respectively after the first 174, 346 and 518 patients enrolled have completed the 90-day follow-up. The interval may be more frequent if requested by the Data and Safety Monitoring Board (DSMB). At interim analysis, in case the stopping boundaries are crossed the DSMB may recommend stopping the study either for better efficacy of the tested treatment either for futility. Other factors, such as safety, will be taken into consideration by the DSMB in the decision to stop the study. When considering stopping the trial for safety reasons, the DSMB will be instructed to consider both mortality (mRS=6) and severe dependency (mRS=5) at 3 months as one single outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke where patient is ineligible for IV thrombolytic treatment or the treatment is contraindicated (e.g., subject presents beyond recommended time from symptom onset), or where patient has received IV thrombolytic therapy without clinical improvement.
2. No significant pre-stroke functional disability (mRS ≤ 1)
3. Baseline NIHSS score obtained prior to randomization must be equal or higher than 8 points
4. Age ≥18 years
5. Occlusion (TICI 0-1) of the intracranial ICA (distal ICA or T occlusions) and/or MCA-M1 segment suitable for endovascular treatment, as evidenced by CTA, MRA or angiogram, with or without concomitant cervical carotid occlusion or stenosis.
6. Patient treatable within eight hours of symptom onset. Symptoms onset is defined as point in time the patient was last seen well (at baseline). Treatment start is defined as groin puncture.
7. Informed consent obtained from patient or acceptable patient surrogate

Exclusion Criteria:

1. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0
2. Baseline platelet count < 30.000/µL
3. Baseline blood glucose of < 50mg/dL or > 400mg/dl
4. Severe, sustained hypertension (SBP > 185 mm Hg or DBP > 110 mm Hg) NOTE: If the blood pressure can be successfully reduced and maintained at the acceptable level using AHA guidelines recommended medication (including iv antihypertensive drips), the patient can be enrolled.
5. Patients in coma (NIHSS item of consciousness >1) (Intubated patients for transfer could be randomized only in case an NIHSS is obtained by a neurologist prior transportation).
6. Seizures at stroke onset which would preclude obtaining a baseline NIHSS
7. Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
8. History of life threatening allergy (more than rash) to contrast medium
9. Subjects who has received IV t-PA treatment beyond 4,5 hours from the beginning of the symptoms
10. Woman of childbearing potential who is known to be pregnant or lactating or who has a positive pregnancy test on admission.
11. Subject participating in a study involving an investigational drug or device that would impact this study.
12. Cerebral vasculitis
13. Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, mRS score at baseline must be ≤1. This excludes patients who are severely demented, require constant assistance in a nursing home type setting or who live at home but are not fully independent in activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.)
14. Unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitor from overseas).
15. Hypodensity on CT or restricted diffusion amounting to an ASPECTS score of <6 on NCCT, or <5 on DWI MRI. The use of CTP or MRI perfusion is optional.
16. Collaterals with malignant profile on CTA (without colateral circulation on CTA)
17. CT or MR evidence of hemorrhage (the presence of GRE microbleeds is allowed).
18. Significant mass effect with midline shift.
19. Evidence of ipsilateral carotid occlusion, high grade stenosis or arterial dissection in the extracranial or petrous segment of the internal carotid artery that cannot be treated or will prevent access to the intracranial clot or excessive tortuosity of cervical vessels precluding device delivery/deployment
20. Subjects with occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation)
21. Evidence of intracranial tumor (except small meningioma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Distribution of the modified Rankin Scale scores (shift analysis) | 90 days
  Distribution of the modified Rankin Scale scores at 90 days (shift analysis) as evaluated by two separate assessors who are blinded to treatment

SECONDARY OUTCOMES:
Functional independence (modified Rankin Score ≤ 2) | 90 days
  Functional independence measured by modified Rankin Score ≤ 2 in 90 days in both groups
Infarct Burden at 24 hours | 24 hours
  ASPECTS change from baseline to 24 hours on CT or MRI
Dramatic early favorable response | 24 hours
  defined as an NIHSS score 0-2 or a NIHSS score decrease of ≥8 from baseline at 24 hours
Cost effectiveness | Life-time horizon perspective
  Cost effectiveness analysis of interventional therapy vs medical therapy alone
Quality of life analysis | 3 months, 6 months, 1 year
  Quality of life analysis as measured by EuroQol/EQ5D at 3 month, 6 months and one year, between interventional therapy vs medical therapy alone
Vessel recanalization at 24 hours | 24 hours
  Vessel recanalization evaluated by CT angiography (CTA) or MR angiography (MRA) at 24 hours in both treatment groups
Successful recanalization at the end of procedure | immediatelly after procedure (only thrombectomy arm)
  defined as a grade of 2b or 3 (indicating reperfusion of >50% of the affected territory) on the modified Thrombolysis in Cerebral Infarction (mTICI) scale
Mortality | 90 days
  Mortality at 90 days
Symptomatic Intracranial hemorrhage | 24 hours
  Clinically significant Intracranial hemorrhage (ICH) rates at 24 (-2/+12) hours. All intracerebral hemorrhages will be classified by a central core-lab using the ECASS criteria for CT evaluation. Symptomatic ICH will be defined as per the SITS-MOST definition: deterioration in NIHSS score of ≥4 points within 24 hours from treatment and evidence of intraparenchymal hemorrhage type 2 in the 22 to 36 hours follow-up imaging scans. The incidence of any asymptomatic hemorrhage measured at 24 (-2/+12) hours will also be compared
Procedure related complications | During the procedure
  Complications occurring during the procedure will be evaluated: distal embolization in a new territory, arterial dissection, arterial perfuration, groin hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Raul Nogueira, MD, Principal Investigator — Emory University; Sheila CO Martins, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (15):
- Brazil (15):
  - Hospital Geral de Fortaleza/SUS, Fortaleza, Ceará
  - Hospital Estadual Central, Vitória, Espírito Santo
  - Hospital Geral Roberto Santos, Salvador, Estado de Bahia
  - Hospital de Base do Distrito Federal, Brasília, Federal District
  - Hospital de Clínicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Hospital São José do Avaí, Itaperuna, Rio de Janeiro
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UNIÃO BRASILEIRA DE EDUCAÇÃO E ASSISTENCIA, Hospital São Lucas PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Governador Celso Ramos, Florianópolis, Santa Catarina
  - Clinica Neurologica e Neurocirurgica de Joinville S/S Ltda, Joinville, Santa Catarina
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - Hospital de Clínicas - UNICAMP, Campinas, São Paulo
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Irmandade da Santa Casa de Misericórdia, São Paulo, São Paulo
  - Universidade Federal de São Paulo - UNIFESP/EPM, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva GS, Alves MM, Barros FCD, Frudit ME, Pontes-Neto OM, Mont'Alverne FJ, Rebello LC, Carbonera LA, Abud DG, Lima F, de Souza AC, Liebeskind D, Mosmann G, Bezerra D, Saver J, Cardoso F, Nogueira RG, Martins SO. The role of intravenous thrombolysis before mechanical Thrombectomy: A subgroup analysis of the RESILIENT trial. J Neurol Sci. 2024 Feb 15;457:122853. doi: 10.1016/j.jns.2023.122853. Epub 2023 Dec 20. PMID 38182456
- [Derived] Martins SO, Mont'Alverne F, Rebello LC, Abud DG, Silva GS, Lima FO, Parente BSM, Nakiri GS, Faria MB, Frudit ME, de Carvalho JJF, Waihrich E, Fiorot JA Jr, Cardoso FB, Hidalgo RCT, Zetola VF, Carvalho FM, de Souza AC, Dias FA, Bandeira D, Miranda Alves M, Wagner MB, Carbonera LA, Oliveira-Filho J, Bezerra DC, Liebeskind DS, Broderick J, Molina CA, Fogolin Passos JE, Saver JL, Pontes-Neto OM, Nogueira RG; RESILIENT Investigators. Thrombectomy for Stroke in the Public Health Care System of Brazil. N Engl J Med. 2020 Jun 11;382(24):2316-2326. doi: 10.1056/NEJMoa2000120. PMID 32521133
- [Derived] Gagliardi VDB, Gagliardi RJ. Current and future conditions of stroke care in Brazil. Arq Neuropsiquiatr. 2019 Jan;77(1):68-69. doi: 10.1590/0004-282X20180160. No abstract available. PMID 30758449